CLINICAL TRIAL: NCT02950545
Title: Evaluating and Improving Functional Driving Vision of Patients With Astigmatism: Phase 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Cox, PhD, Professor, Departments of Psychiatry, Internal Medicine and Ophthalmology, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18499
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Astigmatism
Keywords: astigmatism, contact lens, driving
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo, Spherical, then Toric Lenses (Experimental): Crossover order 1
  Interventions: Device: Placebo Lenses; Device: Spherical Lenses; Device: Toric Lenses
- Placebo, Toric, then Spherical Lenses (Experimental): Crossover order 2
  Interventions: Device: Placebo Lenses; Device: Spherical Lenses; Device: Toric Lenses
- Spherical, Placebo, then Toric Lenses (Experimental): Crossover order 3
  Interventions: Device: Placebo Lenses; Device: Spherical Lenses; Device: Toric Lenses
- Spherical, Toric, then Placebo Lenses (Experimental): Crossover order 4
  Interventions: Device: Placebo Lenses; Device: Spherical Lenses; Device: Toric Lenses
- Toric, Placebo, then Spherical Lenses (Experimental): Crossover order 5
  Interventions: Device: Placebo Lenses; Device: Spherical Lenses; Device: Toric Lenses
- Toric, Spherical, then Placebo Lenses (Experimental): Crossover order 6
  Interventions: Device: Placebo Lenses; Device: Spherical Lenses; Device: Toric Lenses

INTERVENTIONS:
Device: Placebo Lenses — AcuVue Oasys Bandage Lenses with no prescription
Device: Spherical Lenses — 1-DAY ACUVUE® MOIST contact lenses
Device: Toric Lenses — 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses

SUMMARY:
It is a common clinical practice to leave small amounts of astigmatism uncorrected in contact lens wearers. Therefore, some drivers who have astigmatism and wear contact lenses may experience blur while driving. The purpose of this study is to determine if correcting small amounts of astigmatism with contact lenses will improve driving safety.

DETAILED DESCRIPTION:
The purpose of this randomized control trial is to compare visual performance and simulated driving performance of adults with astigmatism when wearing 1*DAY ACUVUE® MOIST for ASTIGMATISM (toric), 1*DAY ACUVUE® MOIST (spherical control), and 1*DAY ACUVUE® MOIST (placebo) contact lenses. Adult subjects with nearsightedness and astigmatism will wear three types of soft contact lenses (placebo, spherical and toric in randomized order). Each subject will read letters on standard eye charts and complete vision and driving tests in a driving simulator. Subjects will repeat these tests with each lens type. Analyses will include an ANOVA to look for a main effect of lens condition, and separate contrasts to compare toric vs. spherical, toric vs. placebo, and spherical vs. placebo lenses. Investigating the lenses under simulated driving conditions, which involve eye movement demands, will lend insight into the potential advantages of toric over spherical contact lenses for driving safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult licensed driver
* Ages 18-39 years
* Corrected vision of 20/40 or better in each eye
* Astigmatism between 0.75 and 1.75 diopters in each eye
* Nearsightedness between 0 and -9 diopters in each eye
* No active eye infection
* No defective peripheral vision
* No bifocal correction
* Routinely wears toric contact lenses (more than 4 times per week)
* Routinely drives a car (more than 4 times per week)
* No history of motion, sea, or big screen (e.g. IMAX) sickness, and no persistent Simulation Adaptation Syndrome

Exclusion Criteria:

* Corrected vision worse than 20/40 in either eye
* No astigmatism in either eye
* Active eye infection
* Defective peripheral vision
* Wears bifocals
* Wears contact lenses less than 4 times per week
* Drives infrequently (less than 4 times per week)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Driving Safety Laboratory, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and protocol will be shared on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available on request
Access Criteria: data will be shared via e-mail.

REFERENCES:
- [Background] Cox DJ, Banton T, Record S, Grabman JH, Hawkins RJ. Does correcting astigmatism with toric lenses improve driving performance? Optom Vis Sci. 2015 Apr;92(4):404-11. doi: 10.1097/OPX.0000000000000554. PMID 25946099

RESULTS

PARTICIPANT FLOW:
Groups:
- Crossover Order 1: Placebo, Spherical, then Toric lenses
- Crossover Order 2: Placebo, Toric, then Spherical lenses
- Crossover Order 3: Spherical, Placebo, then Toric lenses
- Crossover Order 4: Spherical, Toric, then Placebo lenses
- Crossover Order 5: Toric, Placebo, then Spherical lenses
- Crossover Order 6: Toric, Spherical, then Placebo lenses
Period: Session 1 (70 Minutes)
Arm/Group | Crossover Order 1 | Crossover Order 2 | Crossover Order 3 | Crossover Order 4 | Crossover Order 5 | Crossover Order 6
Started | 9 | 9 | 7 | 8 | 8 | 10
Completed | 9 | 9 | 7 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout 1 (5 Minutes)
Arm/Group | Crossover Order 1 | Crossover Order 2 | Crossover Order 3 | Crossover Order 4 | Crossover Order 5 | Crossover Order 6
Started | 9 | 9 | 7 | 8 | 8 | 9
Completed | 8 | 9 | 7 | 7 | 8 | 8
Not Completed | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 1
Period: Session 2 (70 Minutes)
Arm/Group | Crossover Order 1 | Crossover Order 2 | Crossover Order 3 | Crossover Order 4 | Crossover Order 5 | Crossover Order 6
Started | 8 | 9 | 7 | 7 | 8 | 8
Completed | 8 | 9 | 7 | 7 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout 2 (5 Minutes)
Arm/Group | Crossover Order 1 | Crossover Order 2 | Crossover Order 3 | Crossover Order 4 | Crossover Order 5 | Crossover Order 6
Started | 8 | 9 | 7 | 7 | 7 | 8
Completed | 7 | 9 | 7 | 7 | 7 | 8
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Session 3 (70 Minutes)
Arm/Group | Crossover Order 1 | Crossover Order 2 | Crossover Order 3 | Crossover Order 4 | Crossover Order 5 | Crossover Order 6
Started | 7 | 9 | 7 | 7 | 7 | 8
Completed | 7 | 9 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover Order 1 | Crossover Order 2 | Crossover Order 3 | Crossover Order 4 | Crossover Order 5 | Crossover Order 6 | Total
Number analyzed (Participants) | 9 | 9 | 7 | 8 | 8 | 10 | 51
Age, Categorical [Count of Participants; unit: Participants] — Participants were 18 to 39 years old
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 9 | 9 | 7 | 8 | 8 | 10 | 51
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 4 | 6 | 7 | 8 | 36
  Male | 5 | 2 | 3 | 2 | 1 | 2 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 7 | 8 | 8 | 10 | 51
Tactical composite [Mean (Standard Deviation); unit: sum of z scores] — This scale measures driving performance in the simulator. It is the sum of the z scores from 15 different driving simulator variables related to braking, steering, speed control and judgment. The scale has no fixed limits. A score of 0 indicates average performance. Higher scores indicate better performance. Population: Only subjects who completed all 3 lens conditions were analyzed. Nine were not analyzed due to study withdrawal (7), receiving the wrong contact lens prescription (1), and having missing data.(1).
  sum of z scores
    Placebo Lenses: number analyzed (Participants) | 7 | 8 | 7 | 7 | 7 | 6 | 42
    Placebo Lenses | -8.93 (6.42) | -4.94 (3.00) | 5.32 (1.77) | 3.32 (3.49) | -0.58 (5.77) | 2.80 (2.82) | -0.69 (6.44)
    Spherical Lenses: number analyzed (Participants) | 7 | 8 | 7 | 7 | 7 | 6 | 42
    Spherical Lenses | 0.99 (6.27) | 2.26 (5.66) | -2.59 (3.24) | -4.67 (4.73) | 3.53 (3.39) | 2.78 (1.81) | 0.37 (5.22)
    Toric Lenses: number analyzed (Participants) | 7 | 8 | 7 | 7 | 7 | 6 | 42
    Toric Lenses | 1.92 (5.00) | 1.88 (3.51) | 5.32 (3.16) | 3.71 (2.66) | -5.18 (4.55) | -7.03 (6.06) | 0.32 (6.00)
Operational composite [Mean (Standard Deviation); unit: sum of z scores] — This scale measures driving-relevant visual performance. It is the sum of the z scores from 5 different driving simulator variables related to visual testing done in the simulator. The scale has no fixed limits. A score of 0 indicates average performance. Higher scores indicate better performance. Population: Only subjects who completed all 3 lens conditions were analyzed. Nine were not analyzed due to study withdrawal (7), receiving the wrong contact lens prescription (1), and having missing data.(1).
  sum of z scores
    Placebo lenses: number analyzed (Participants) | 7 | 8 | 7 | 7 | 7 | 6 | 42
    Placebo lenses | -3.95 (3.95) | -4.91 (4.15) | -2.85 (3.23) | -0.78 (4.51) | -7.43 (4.36) | -4.40 (6.28) | -4.06 (4.64)
    Spherical lenses: number analyzed (Participants) | 7 | 8 | 7 | 7 | 7 | 6 | 42
    Spherical lenses | 1.28 (1.32) | 1.76 (1.27) | 1.61 (0.60) | 3.15 (1.12) | 2.70 (0.74) | 1.52 (1.39) | 2.01 (1.25)
    Toric lenses: number analyzed (Participants) | 7 | 8 | 7 | 7 | 7 | 6 | 42
    Toric lenses | 2.29 (1.16) | 1.70 (1.08) | 3.01 (2.01) | 2.45 (1.53) | 1.30 (0.44) | 1.56 (1.99) | 2.05 (1.48)

OUTCOME MEASURES:

1. Primary Outcome: Tactical Composite Score
Description: This scale measures driving performance in the simulator. It is the sum of the z scores from 15 different driving simulator variables related to braking, steering, speed control and judgment. The scale has no fixed limits. A score of 0 indicates average performance. Higher scores indicate better performance.
Time Frame: 1 day
Population: All participants who completed the 3 simulated driving sessions and who had complete and accurate data records were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Study Participants: Each participant completed (1) Simulated driving with Placebo Lenses (AcuVue Oasys Bandage Lenses with no prescription), (2) Simulated driving with Spherical Lenses (1-DAY ACUVUE® MOIST contact lenses), (3) Simulated driving with Toric Lenses (1-DAY ACUVUE® MOIST for ASTIGMATISM contact...
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
score on a scale
  Placebo | 0.34 (2.44)
  Sphere | -0.01 (2.65)
  Toric | -0.33 (2.77)

2. Secondary Outcome: Operational Composite Score
Description: This scale measures driving-relevant visual performance. It is the sum of the z scores from 5 different driving simulator variables related to visual testing done in the simulator. The scale has no fixed limits. A score of 0 indicates average performance. Higher scores indicate better performance.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
score on a scale
  Placebo | -4.06 (4.64)
  Sphere | 2.01 (1.25)
  Toric | 2.05 (1.48)

ADVERSE EVENTS:
Time Frame: 10 months
Groups:
- Placebo: Participants wore the placebo contact lenses during testing
- Spherical: Participants wore the spherical contact lenses during testing
- Toric: Participants wore the toric contact lenses during testing
Arm/Group | Placebo | Spherical | Toric
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 2/51 | 2/51 | 3/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Spherical (N=51) | Toric (N=51)
Simulation sickness (General disorders) | 2 | 2 | 3 — motion sickness induced by simulator use.

LIMITATIONS AND CAVEATS:
The study primarily investigated vehicle control. Object recognition is also a critical aspect of driving, but was not fully investigated in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT02950545/Prot_SAP_000.pdf